CLINICAL TRIAL: NCT06386900
Title: The Impact of Grand Tour Cyling on Sleep and the Hematological and Metabolomic Profile in World-class Cyclists
Brief Title: The Impact of Grand Tour Cycling on Sleep and the Hematological and Metabolomic Profile in World-class Cyclists
Status: Enrolling by invitation | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Chiel Poffé, Principal investigator, KU Leuven
Other Study IDs: S67595
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Overreaching
Keywords: Cycling; Grand Tour; Sleep; Metabolomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Whole blood
  * Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite cyclists participating in a Grand Tour: * Sleep metrics will be tracked by a smart ring (OURA Gen3, OURA Health Ltd, Oulu, Finland) starting from one month prior to the start till the end of the Grand Tour
  * Nocturnal heart rate and heart rate variability will be collected by a smart ring (OURA Gen3, OURA Health Ltd, Oulu, Finland) starting from one month prior till the end of the Grand Tour
  * Fasted whole blood samples and urine samples will be collected on the morning of (i) the first stage, (ii) the first restday, (iii) second restday, and (iv) last stage of the GrandTour (only in one Grand Tour for a total of 8 cyclists).
  Interventions: Other: Cyclist

INTERVENTIONS:
Other: Cyclist — Participating in the Grand Tour as cyclist

SUMMARY:
This project aims to identify the effect of a 3-week Grand Tour (e.g. Tour de France, Giro d'Italia, and Vuelta a España) on sleep, hematological parameters and the serum metabolome in world-class cyclists.

ELIGIBILITY:
Inclusion Criteria:

* Cylist participating in a Grand Tour (e.g. Tour de France, Vuelta a España, Giro d'Italia)

Exclusion Criteria:

* /

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: Elite cyclist participating in a Grand Tour (e.g. Tour de France, Vuelta a España, Giro d'Italia)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum metabolome abundance of cyclists participating in a Grand Tour | Start of the Grand Tour - restday 1 of the Grand Tour - restday 2 of the Grand Tour - last day of the Grand Tour
  Changes in the abundance of serum metabolites within the cyclists between 4 timepoints (measured by mass spectrometry)
Sleep efficiency during the Grand Tour | Every night starting from one week before till the last night of the Grand Tour
  Percentage change in sleep efficiency during the Grand Tour (measured by OURA ring)
Total sleep time during the Grand Tour | Every night starting from one week before till the last night of the Grand Tour
  Change in total sleep time during the Grand Tour (measured by OURA ring)
Blood haemoglobin concentration | Start of the Grand Tour - restday 1 of the Grand Tour - restday 2 of the Grand Tour - last day of the Grand Tour
  Change in the blood haemoglobin concentration during the Grand Tour

SECONDARY OUTCOMES:
Wakefulness after sleep onset | Every night starting from one week before till the last night of the Grand Tour
  Percentage change in wakefulness after sleep onset during the Grand Tour (measured by OURA ring)
Light sleep | Before the start of the Tour - restday 1 - restday 2 - end of Grand Tour
  Percentage change in light sleep during the Grand Tour (measured by OURA ring)
Deep sleep | Before the start of the Tour - restday 1 - restday 2 - end of Grand Tour
  Percentage change in deep sleep during the Grand Tour (measured by OURA ring)
REM sleep | Before the start of the Tour - restday 1 - restday 2 - end of Grand Tour
  Percentage change in REM sleep during the Grand Tour (measured by OURA ring)
Red blood cell concentration | Start of the Grand Tour - restday 1 of the Grand Tour - restday 2 of the Grand Tour - last day of the Grand Tour
  Change in red blood cell concentration during the Grand Tour
Subjective fatigue | Start of the Grand Tour - restday 1 of the Grand Tour - restday 2 of the Grand Tour - last day of the Grand Tour
  Absolute change in subjective fatigue during the Grand Tour (measured by 11-point scale)

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No